CLINICAL TRIAL: NCT00567554
Title: A Phase III Trials Program Exploring the Integration of Bevacizumab, Everolimus (RAD001), and Lapatinib Into Current Neoadjuvant Chemotherapy Regimes for Primary Breast Cancer
Brief Title: Bevacizumab, Everolimus (RAD001), and Lapatinib as Neoadjuvant Chemotherapy Regimes for Primary Breast Cancer
Acronym: GeparQuinto
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GBG Forschungs GmbH (Other)
Collaborators: AGO Study Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GBG 44; 2006-005834-19 (EudraCT Number)
Record Dates: First submitted 2007-12-04; First posted 2007-12-05 (Estimated); Last update posted 2016-02-10 (Estimated); Status verified 2016-02

CONDITIONS: Breast Cancer
Keywords: breast cancer; primary systemic therapy; pCR Rates; Bevacizumab; Trastuzumab; Lapatinib; Everolimus
MeSH Terms: conditions — Breast Neoplasms | interventions — EC regimen; Docetaxel; Bevacizumab; Paclitaxel; Everolimus; Trastuzumab; Lapatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- 1 (Experimental): EC-T
  Interventions: Drug: epirubicin - cyclophosphamide / docetaxel
- 2 (Experimental): EC-T +/- B
  Interventions: Drug: epirubicin - cyclophosphamide / docetaxel + bevacizumab
- 3 (Experimental): Pw
  Interventions: Drug: paclitaxel
- 4 (Experimental): Pw + RAD001
  Interventions: Drug: paclitaxel + everolimus (RAD001)
- 5 (Experimental): EC-T + H
  Interventions: Drug: epirubicin - cyclophosphamide / docetaxel + trastuzumab
- 6 (Experimental): EC-T + L
  Interventions: Drug: epirubicin - cyclophosphamide / docetaxel + lapatinib

INTERVENTIONS:
Drug: epirubicin - cyclophosphamide / docetaxel
  Arms: 1
Drug: epirubicin - cyclophosphamide / docetaxel + bevacizumab
  Arms: 2
Drug: paclitaxel
  Arms: 3
Drug: paclitaxel + everolimus (RAD001)
  Arms: 4
Drug: epirubicin - cyclophosphamide / docetaxel + trastuzumab
  Arms: 5
Drug: epirubicin - cyclophosphamide / docetaxel + lapatinib
  Arms: 6

SUMMARY:
Anthracycline-taxane based chemotherapy regimens are recommended mainly by current guidelines for neoadjuvant application of systemic treatment. The addition of other cytotoxic agents, e.g. antimetabolites, vincaalkaloids, or platinum salts resulted in marginal increase in efficacy, but was associated also with an increase in toxicity. Recently, only the addition of the Her-2 antibody trastuzumab has significantly improved pathologic response rate.

Therefore, two major strategies are followed in current research projects:

* To improve the selection of patients according to their tumors' sensitivity to chemotherapy.
* To implement small molecules with specific mechanism of action.

Within the GeparQuinto trial, the first strategy is followed by:

* The PREDICT substudy. A gene signature specific for the response to anthracyclines and taxanes will be prospectively evaluated for its ability to identify patients with chance higher than 50% for a pCR. The results may leed to a better risk-benefit ratio for the use of conventional chemotherapy.
* Adapting further chemotherapy to the response of the tumor to the first couple of chemotherapy cycles. Based on the previous experience made by the GeparTrio study, patients not responding early have a low chance to respond with a pCR irrespective of the type of chemotherapy. So, if further chemotherapy is planned, therapy should be selected according to a favorable toxicity profile.

The second strategy is followed by investigating in three parallel group comparisons the efficiency of three distinct small molecules which appear to be generally active in breast cancer:

* Bevacizumab, an inhibitor of the VEGF pathway targeting tumor neo-angiogenesis.
* Lapatinib, an inhibitor of the Her-1 and Her-2 receptor tyrosine kinase.
* RAD001 (Everolimus), an inhibitor of the mTOR molecule, a central controller of tumor cell growth and angiogenesis and chemosensitizer.

Treatment for patients participating in the GeparQuinto study will be allocated according to the Her-2 status of the tumor as well as according to the sonographic response after the first 4 cycles of treatment. Experimental therapy with bevacizumab, lapatinib, and everolimus (RAD001) will be randomly added in distinct settings.

DETAILED DESCRIPTION:
Primary objectives:

To compare the pCR rates of neoadjuvant treatment of epirubicin / cyclophosphamide followed by docetaxel (EC-T) with or without bevacizumab (EC-T vs. ECB-TB) in patients with Her-2 negative primary breast cancer (Setting I).

To compare the pCR rates of neoadjuvant treatment with weekly paclitaxel with or without Everolimus (RAD001) (Pw vs. PwR) in patients with Her-2 negative primary breast cancer showing no sonographic response to 4 cycles of EC +/-B (Setting II).

To compare the pCR rates of neoadjuvant treatment with epirubicin / cyclophosphamide followed by docetaxel with either trastuzumab or lapatinib (ECH-TH vs. ECL-TL) in patients with Her-2 positive primary breast cancer (Setting III).

Secondary objectives:

1. To assess the toxicity of and compliance to all six treatments.
2. To determine the response rates of the breast tumor and axillary nodes by physical examination and imaging tests (sonography, mammography, or MRI) after treatment in all arms.
3. To determine the breast conservation rate after each treatment.
4. To determine the (loco-regional and distant) disease-free and overall survival after each treatment. In Her-2 positive disease, the cerebral disease-free survival will be determined separately.
5. To assess treatment efficacies in subgroups defined according to tumor stage (T2-3 vs. T4), receptor status (ER and / or PgR positive vs. ER and PgR negative) and response by best appropriate imaging method to the first four cycles of treatment (complete vs. partial vs. no change).
6. To examine and compare pre-specified molecular markers such as Ki-67, phospho-mTOR, YB-1, COX-2, HuR, phospho-p70 S6K, p65 NF kappa B, PTEN, PI3-K, Akt, and a marker for stem cell like breast cancers (SOX-10) on core biopsy before and after end of chemotherapy.

Objectives of Substudies:

1. To assess and correlate circulating tumor cells and proteins with the effect of treatment(CTC Substudy).
2. To compare the pathologic complete response (pCR), breast conservation, clinical and imaging response rate (after four cycles and before surgery) in patients where the tumor shows a favorable profile of a predetermined combined biomarker set to those where the tumor does not show it (PREDICT Substudy).
3. To determine the percentage of patients in which conventional axillary clearance can be substituted by sentinel node biopsy when a predetermined clinical algorithm is used (SENTINA Substudy).
4. To assess the surgical outcome according to patient's and surgeon's perspectives in correlation with clinical and pathological response to systemic treatment (SOS - Surgical Outcome Substudy).
5. To correlate Single Nucleotide Polymorphisms (SNPs) of genes which are either involved in the metabolism or in the effectiveness of the distinct therapies with the associated toxicity and histologically assessed treatment effect (Pharmacogenomic Substudy).

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. Complete baseline documentation sent to GBG Forschungs GmbH;
3. Unilateral or bilateral primary carcinoma of the breast, confirmed histologically by core biopsy. Fine-needle aspiration is not sufficient. Incisional biopsy is not allowed.
4. Tumor lesion in the breast with a palpable size of ≥ 2 cm or a sonographically size of at least 1 cm in maximum diameter. The lesion has to be measurable in two-dimensions preferably by sonography. In case of inflammatory disease the extent of inflammation can be used as measurable lesion;
5. Patients should have stages of disease in which adjuvant chemotherapy would be considered.

   * Locally advanced tumors with cT4 or cT3 or
   * Estrogen (ER)- and progesterone (PgR)-receptor negative tumors or
   * ER or PgR positive tumors which are cN+ (for cT2) or pNSLN+ (for cT1) * During the Run-In-Safety phase only patients with cT4 or cT3 cN+ disease are eligible.
6. Known HER-2/neu status detected on core biopsy. HER-2/neu positive is defined as HercepTest IHC 3+ or FISH+;
7. Age older than 18 years;
8. Karnofsky Performance status index at least 80%;
9. Normal cardiac function must be confirmed by ECG and cardiac ultrasound (LVEF or shortening fraction) within 1 month prior to registration.
10. Laboratory requirements:

    Hematology: Absolute neutrophil count (ANC) ≥ 2.0 x 10e9/L platelets ≥ 100 x 10e9/L, Hemoglobin ≥ 10 g/dL (≥ 6.2 mmol/L) Hepatic function: Total bilirubin < 1 x UNL ASAT (SGOT) and ALAT (SGPT)≤ 2.5 x UNL Alkaline phosphatase ≤ 5 UNL. Patients with ASAT and / or ALAT > 1.5 x UNL associated with alkaline phosphatase > 2.5 x UNL are not eligible for the study; Renal function: Creatinine ≤ 175 µmol/L (2 mg/dL) < 1,25 UNL (or the calculated creatinine clearance ≥ 60 mL/min) Urine dipstick for proteinuria < 2+. Patients discovered to have ≥2+ proteinuria on dipstick urinalysis should undergo a 24 hour urine collection and must demonstrate ≤1 g of protein in 24 hours
11. Paraffin tumor tissue block and two serum samples centrally made available
12. Negative pregnancy test (urine or serum)
13. Complete staging work-up within 3 months prior to registration.
14. Patients must be available and compliant for treatment and follow-up.

Exclusion criteria:

1. Patients with low or moderate risk, which are only doubtful candidates for adjuvant chemotherapy
2. Evidence of distant metastasis;
3. Prior chemotherapy for any malignancy;
4. Prior radiation therapy for breast cancer;
5. Pregnant or lactating patients.
6. Inadequate general condition
7. Previous malignant disease
8. Known or suspected congestive heart failure (>NYHA I) and/or coronary heart disease, angina pectoris requiring antianginal medication, previous history of myocardial infarction, evidence of transmural infarction on ECG, un- or poorly controlled arterial hypertension, rhythm abnormalities requiring permanent treatment, clinically significant valvular heart disease
9. Previous thromboembolic event
10. Known hemorrhagic diathesis or increased bleeding risk
11. History of significant neurological or psychiatric disorders that would prohibit the understanding and giving of informed consent;
12. Pre-existing motor or sensory neuropathy of a severity more than grade 2 by NCI criteria
13. Currently active infection;incomplete wound healing
14. Active peptic ulcer
15. Disease significantly affecting gastrointestinal function
16. History of abdominal fistula, gastrointestinal perforation or intra-abdominal abscess within 6 months of enrollment
17. Severe pulmonary condition/illness
18. Unstable diabetes mellitus; insulin dependent type II diabetes mellitus
19. Major surgery or incomplete wound healing within the last 28 days
20. Definite contraindications for the use of corticosteroids
21. Known hypersensitivity reaction to one of the investigational compounds or incorporated substances; or known dihydropyrimidine dehydrogenase deficiency
22. Concurrent treatment with:chronic corticosteroids unless initiated > 6 months prior to study entry and at low dose (20 mg methylprednisolone or equivalent); sex hormones.Virostatic agents like sorivudine or analogs like brivudine, concurrent treatment with aminoglycosides; anticoagulants: heparin, warfarin as well as acetic acid (e.g. Aspirin®) at a dose of > 325mg/day or clopidogrel at a dose of > 75 mg/day)e.other experimental drugs or any other anti-cancer therapy; drugs recognized as being strong inhibitors or inducers of the isoenzyme CYP3A (e.g. Rifabutin, Rifampicin, Clarithromycin, Ketoconazole, Itraconazole, Ritonavir, Telithromycin, Erythromycin, Verapamil, Dilitazem, within the last 5 days or the expected need for these treatments during study participation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2600 (Actual)
Dates: Start 2007-10; Primary Completion 2011-08 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
To compare the pCR rates of neoadjuvant treatment in all 3 Settings | 2009

SECONDARY OUTCOMES:
To assess the toxicity of and compliance to all six treatments. | 2009
To determine the breast conservation rate after each treatment. | 2009
To determine the (loco-regional and distant) disease-free and overall survival after each treatment. In Her-2 positive disease the cerebral disease-free survival will be determined separately. | 2012
To assess treatment efficacies in subgroups defined according to tumor stage (T2-3 vs T4) receptor status (ER and/or PR pos. vs ER and PR neg.) and response by best appropriate imaging method to the first 4 cycles of treatment (complete vs partial vs no) | 2009
To examine and compare prespecified molecular markers on core biopsy before and after end of chemotherapy | 2012

CONTACTS AND LOCATIONS:
Overall Officials: Gunter von Minckwitz, MD, Prof., Principal Investigator — GBG Forschungs GmbH; Michael Untch, MD, Prof., Study Chair — AGO Study Group
Locations (1):
- Universitätsfrauenklinik Frankfurt / Main, Frankfurt am Main, Germany

REFERENCES:
- [Derived] Fasching PA, Loibl S, Hu C, Hart SN, Shimelis H, Moore R, Schem C, Tesch H, Untch M, Hilfrich J, Rezai M, Gerber B, Costa SD, Blohmer JU, Fehm T, Huober J, Liedtke C, Weinshilboum RM, Wang L, Ingle JN, Muller V, Nekljudova V, Weber KE, Rack B, Rubner M, von Minckwitz G, Couch FJ. BRCA1/2 Mutations and Bevacizumab in the Neoadjuvant Treatment of Breast Cancer: Response and Prognosis Results in Patients With Triple-Negative Breast Cancer From the GeparQuinto Study. J Clin Oncol. 2018 Aug 1;36(22):2281-2287. doi: 10.1200/JCO.2017.77.2285. Epub 2018 May 23. PMID 29791287
- [Derived] Untch M, von Minckwitz G, Gerber B, Schem C, Rezai M, Fasching PA, Tesch H, Eggemann H, Hanusch C, Huober J, Solbach C, Jackisch C, Kunz G, Blohmer JU, Hauschild M, Fehm T, Nekljudova V, Loibl S; GBG and the AGO-B Study Group. Survival Analysis After Neoadjuvant Chemotherapy With Trastuzumab or Lapatinib in Patients With Human Epidermal Growth Factor Receptor 2-Positive Breast Cancer in the GeparQuinto (G5) Study (GBG 44). J Clin Oncol. 2018 May 1;36(13):1308-1316. doi: 10.1200/JCO.2017.75.9175. Epub 2018 Mar 15. PMID 29543566
- [Derived] von Minckwitz G, Loibl S, Untch M, Eidtmann H, Rezai M, Fasching PA, Tesch H, Eggemann H, Schrader I, Kittel K, Hanusch C, Huober J, Solbach C, Jackisch C, Kunz G, Blohmer JU, Hauschild M, Fehm T, Nekljudova V, Gerber B; GBG/AGO-B study groups; Gnauert K, Heinrich B, Pratz T, Groh U, Tanzer H, Villena C, Tulusan A, Liedtke B, Blohmer JU, Kittel K, Mau C, Potenberg J, Schilling J, Just M, Weiss E, Buckner U, Wolfgarten M, Lorenz R, Doering G, Feidicker S, Krabisch P, Deichert U, Augustin D, Kunz G, Kast K, von Minckwitz G, Nestle-Kramling C, Rezai M, Hoss C, Terhaag J, Fasching P, Staib P, Aktas B, Kuhn T, Khandan F, Mobus V, Solbach C, Tesch H, Stickeler E, Heinrich G, Wagner H, Abdallah A, Dewitz T, Emons G, Belau A, Rethwisch V, Lantzsch T, Thomssen C, Mattner U, Nugent A, Muller V, Noesselt T, Holms F, Muller T, Deuker JU, Schrader I, Strumberg D, Uleer C, Solomayer E, Runnebaum I, Link H, Tome O, Ulmer HU, Conrad B, Feisel-Schwickardi G, Eidtmann H, Schumacher C, Steinmetz T, Bauerfeind I, Kremers S, Langanke D, Kullmer U, Ober A, Fischer D, Kohls A, Weikel W, Bischoff J, Freese K, Schmidt M, Wiest W, Sutterlin M, Dietrich M, Griesshammer M, Burgmann DM, Hanusch C, Rack B, Salat C, Sattler D, Tio J, von Abel E, Christensen B, Burkamp U, Kohne CH, Meinerz W, Grasshoff ST, Decker T, Overkamp F, Thalmann I, Sallmann A, Beck T, Reimer T, Bartzke G, Deryal M, Weigel M, Huober J, Weder P, Steffens CC, Lemster S, Stefek A, Ruhland F, Hofmann M, Schuster J, Simon W, Kronawitter U, Clemens M, Fehm T, Janni W, Latos K, Bauer W, Rossmann A, Bauer L, Lampe D, Heyl V, Hoffmann G, Lorenz-Salehi F, Hackmann J, Schlag R. Survival after neoadjuvant chemotherapy with or without bevacizumab or everolimus for HER2-negative primary breast cancer (GBG 44-GeparQuinto)dagger. Ann Oncol. 2014 Dec;25(12):2363-2372. doi: 10.1093/annonc/mdu455. Epub 2014 Sep 15. PMID 25223482
- [Derived] von Minckwitz G, Eidtmann H, Rezai M, Fasching PA, Tesch H, Eggemann H, Schrader I, Kittel K, Hanusch C, Kreienberg R, Solbach C, Gerber B, Jackisch C, Kunz G, Blohmer JU, Huober J, Hauschild M, Fehm T, Muller BM, Denkert C, Loibl S, Nekljudova V, Untch M; German Breast Group; Arbeitsgemeinschaft Gynakologische Onkologie-Breast Study Groups. Neoadjuvant chemotherapy and bevacizumab for HER2-negative breast cancer. N Engl J Med. 2012 Jan 26;366(4):299-309. doi: 10.1056/NEJMoa1111065. PMID 22276820
- [Derived] Untch M, Loibl S, Bischoff J, Eidtmann H, Kaufmann M, Blohmer JU, Hilfrich J, Strumberg D, Fasching PA, Kreienberg R, Tesch H, Hanusch C, Gerber B, Rezai M, Jackisch C, Huober J, Kuhn T, Nekljudova V, von Minckwitz G; German Breast Group (GBG); Arbeitsgemeinschaft Gynakologische Onkologie-Breast (AGO-B) Study Group. Lapatinib versus trastuzumab in combination with neoadjuvant anthracycline-taxane-based chemotherapy (GeparQuinto, GBG 44): a randomised phase 3 trial. Lancet Oncol. 2012 Feb;13(2):135-44. doi: 10.1016/S1470-2045(11)70397-7. Epub 2012 Jan 17. PMID 22257523